CLINICAL TRIAL: NCT01926691
Title: Predictors for Poststroke Outcomes: the Tel Aviv Brain Acute Stroke Cohort (TABASCO) Study
Brief Title: Predictors for Poststroke Outcomes: Tel Aviv Brain Acute Stroke Cohort Acute Stroke Cohort (TABASCO)
Acronym: TABASCO
Status: Completed | Type: Observational
Sponsor: Eli Sprecher, MD (Other Government)
Collaborators: Tel Aviv University (Other); Hebrew University of Jerusalem (Other); Technische Universität Dresden (Other); University of New Mexico (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, Director of Research and Development, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TABASCO
Record Dates: First submitted 2013-08-18; First posted 2013-08-21 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Stroke; Dementia; Cerebrovascular Disorders; Alzheimer's Disease; Brain Ischemia
Keywords: dementia; poststroke cognitive impairment; inflammation; stress
MeSH Terms: conditions — Stroke; Dementia; Cerebrovascular Disorders; Alzheimer Disease; Brain Ischemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute First-ever Stroke: Patients over 50 years and without pre-stroke dementia, displaying an ischemic first-ever stroke or transient ischemic attack (TIA), onset within the last 72 hours, Israeli residents.

SUMMARY:
Background: Recent studies have demonstrated that even mild stroke survivors experience residual damage, which persists and in fact increases in subsequent years. About 45% of stroke victims remain with different levels of disability. While studies on cognitive impairment and dementia after stroke are receiving increasing clinical attention, the underlying pathophysiology is poorly understood. Identifying the mechanisms involved and recognizing early biomarkers for individual vulnerability, require a multi-modal approach, as the mechanisms involved in cerebrovascular disease and individual trajectories of post-stroke recovery may impact upon each other on various levels.

Aims and Hypothesis: To date there is no single measure that can be used to identify patients who are prone to develop cognitive impairment and other disabilities from those with better recovery prospects.

We hypothesize that data based on biochemical, neuroimaging, genetic and psychological measures can, in aggregate, serve as better predictors for subsequent disability, cognitive and neurological deterioration, and suggest possible interventions.

Design: The TABASCO (Tel-Aviv Brain Acute Stroke Cohort) study, a prospective cohort study aim to recruit about approximately 1125 consecutive first-ever mild-moderate stroke patients. It is designed to evaluate the association between predefined demographic, psychological, inflammatory, biochemical, neuro-imaging and genetic markers, measured during the acute phase, and long-term outcome: subsequent cognitive deterioration, vascular events (including recurrent strokes), falls, affective changes, functional everyday difficulties and mortality.

Discussion: This study is an attempt to comprehensively investigate the long term outcome of mild-moderate strokes. Its prospective design will provide quantitative data on stroke recurrence, the incidence of other vascular events and the evaluation of cognitive, affective and functional decline. Identifying the factors associated with post stroke cognitive and functional decline could potentially yield more effective therapeutic approaches.

The investigators believe that an extensive approach of analyzing the interaction between different risk factors would more accurately predict neurological and cognitive deterioration.

DETAILED DESCRIPTION:
The primary aim of the TABASCO study is to identify predictors of post stroke cognitive decline. A particular focus will be on inflammatory and stress markers, as well as neuroimaging measures.

Eligibility

Participants are recruited from patients admitted to the Department of Emergency Medicine at the Tel-Aviv Sourasky Medical Center (TASMC) within 72 hours of their first-ever acute ischemic stroke or transient ischemic attack (TIA) symptoms onset.

Criteria

Inclusion Criteria:

1. Age ≥ 50 years
2. Israeli residents
3. Acute stroke/TIA that occurred within the last 3 days as defined by:

   acute focal neurological deficit with a total score on the NIH Stroke Scale (NIHSS) <17
4. Written informed consent by patient prior to study participation
5. Willingness to participate in follow-up

Exclusion Criteria:

patients presenting with a primary hemorrhagic stroke (intracerebral or subarachnoid)

1. history of any preceding cerebral vascular event (excluding previous TIA)
2. imminent death or unconscious state
3. patients unlikely to be released from hospital following the qualifying stroke, or have a severe disability after the qualifying stroke which makes follow-up unlikely
4. known malignant disease or other chronic disease with poor prognosis (predicted survival less than two-years)
5. stroke resulting from trauma or invasive procedure
6. patients with a prestroke history consistent with dementia or cognitive impairment before the stroke
7. severe aphasia.

Stroke diagnosis is verified by senior vascular neurologists and baseline demographic and clinical data are collected. Interviews are conducted by trained interviewers at baseline, 3, 6, 12 and 24 months, and yearly thereafter up to 10 years.

Assessments and data collection A senior vascular neurologist conducts a thorough physical examination and reviews the imaging data and medical records of potential participants to determine eligibility. Participants are asked to consent for all study examinations and a signed informed consent is obtained from patients who agree.

Information is collected for the evaluation of co-morbidities at the time of recruitment and throughout the study.

All subjects are prospectively followed at three-, six-, 12 and 24 months from stroke onset and annually thereafter. Approximately three-months after stroke, consenting participants are visited at home by trained occupational therapists.

For subjects who died, the date of death is recorded along with its cause, based on information obtained from the family, medical records, death certificates and data from the government's official civil registry.

Sample size In an attempt to identify a 40% difference in post stroke cognitive decline, we have calculated the required sample size (Ben Assayag E et al,International Journal of Stroke,Vol 7, June 2012, 341-347).

The investigators aim to recruit at least 1125 participants to allow for loss to follow-up, potential clustering effects, missing data and to provide sufficient numbers for multivariate modeling.

Investigators

Principal Investigators:

Natan Bornstein, Prof. Tel Aviv Sourasky Medical Center Amos Korczyn, Prof. Tel Aviv University Einor Ben Assayag, Phd Tel Aviv Sourasky Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Israeli residents
* Acute stroke that occurred within the last 3 days as defined by:
* acute focal neurological deficit, with a total score on the NIH Stroke Scale (NIHSS) <17
* Written informed consent by patient prior to study participation
* Willingness to participate in follow-up

Exclusion Criteria:

* patients presenting with a primary hemorrhagic stroke (intracerebral or subarachnoid)
* history of any preceding cerebral vascular event (excluding TIA)
* imminent death or unconscious state
* patients unlikely to be released from hospital following the qualifying stroke, or have a severe disability after the
* qualifying stroke which makes follow-up unlikely
* known malignant disease or other chronic disease with poor prognosis (predicted survival less than two-years)
* stroke resulting from trauma or invasive procedure
* patients with a prestroke history consistent with dementia, or cognitive impairment before the stroke
* severe aphasia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Emergency Medicine at the Tel-Aviv Sourasky Medical Center (TASMC) within three-days of their first-ever acute ischemic stroke or transient ischemic attack (TIA) symptoms onset.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
dementia/cognitive decline occurrence | 10 years
  This evaluation will be based on a neurological and general clinical examination, as well as an interview with the patient's family, by a cognitive neurologist, and a senior clinician to determine whether the participant meets the DSM IV criteria for dementia or is defined as minimal cognitive impairment (MCI).

SECONDARY OUTCOMES:
dementia or cognitive decline occurrence | 6 months - 10 years
  Dementia/ cognitive decline occurrence [ Time Frame: 6, 12, 18 months and annually up to 10 years] this evaluation will be based on a neurological and general clinical examination, same as for primary outcome.

OTHER OUTCOMES:
Death or recurrent vascular events occurence | Study entry - 10 years
  Death or recurrent vascular events that occured after the first acute stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Ben Assayag E, Korczyn AD, Giladi N, Goldbourt U, Berliner AS, Shenhar-Tsarfaty S, Kliper E, Hallevi H, Shopin L, Hendler T, Baashat DB, Aizenstein O, Soreq H, Katz N, Solomon Z, Mike A, Usher S, Hausdorff JM, Auriel E, Shapira I, Bornstein NM. Predictors for poststroke outcomes: the Tel Aviv Brain Acute Stroke Cohort (TABASCO) study protocol. Int J Stroke. 2012 Jun;7(4):341-7. doi: 10.1111/j.1747-4949.2011.00652.x. Epub 2011 Nov 2. PMID 22044517
- [Derived] Seyman EE, Sadeh-Gonik U, Berman P, Blum I, Shendler G, Nathan B, Rothschild O, Molad J, Ben Assayag E, Hallevi H; TABASCO prospective cohort study group. Association between intracranial vessel calcifications, structural brain damage, and cognitive impairment after minor strokes: a prospective study. Front Neurol. 2023 Jul 18;14:1218077. doi: 10.3389/fneur.2023.1218077. eCollection 2023. PMID 37533476
- [Derived] Ben Assayag E, Eldor R, Korczyn AD, Kliper E, Shenhar-Tsarfaty S, Tene O, Molad J, Shapira I, Berliner S, Volfson V, Shopin L, Strauss Y, Hallevi H, Bornstein NM, Auriel E. Type 2 Diabetes Mellitus and Impaired Renal Function Are Associated With Brain Alterations and Poststroke Cognitive Decline. Stroke. 2017 Sep;48(9):2368-2374. doi: 10.1161/STROKEAHA.117.017709. Epub 2017 Aug 11. PMID 28801477
- [Derived] Tene O, Shenhar-Tsarfaty S, Korczyn AD, Kliper E, Hallevi H, Shopin L, Auriel E, Mike A, Bornstein NM, Assayag EB. Depressive symptoms following stroke and transient ischemic attack: is it time for a more intensive treatment approach? results from the TABASCO cohort study. J Clin Psychiatry. 2016 May;77(5):673-80. doi: 10.4088/JCP.14m09759. PMID 27035632
- [Derived] Ben Assayag E, Shenhar-Tsarfaty S, Korczyn AD, Kliper E, Hallevi H, Shopin L, Auriel E, Giladi N, Mike A, Halevy A, Weiss A, Mirelman A, Bornstein NM, Hausdorff JM. Gait measures as predictors of poststroke cognitive function: evidence from the TABASCO study. Stroke. 2015 Apr;46(4):1077-83. doi: 10.1161/STROKEAHA.114.007346. Epub 2015 Feb 12. PMID 25677599